CLINICAL TRIAL: NCT02776384
Title: Prognostic and Diagnostic Value of Serial Biomarker Measurements, Echocardiographic Techniques and Cardiopulmonary Function Tests in Patients With Chronic Heart Failure.
Brief Title: Prognostic and Diagnostic Value of Biomarkers and Cardiac Functional Parameters in Patients With Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhang Qi, MD, MD, Shanghai Jiao Tong University School of Medicine
Other Study IDs: RJH-20151127
Record Dates: First submitted 2016-05-15; First posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Heart Failure
Keywords: Heart Failure; Biomarkers; Echocardiography; Cardiopulmonary Function Tests
MeSH Terms: conditions — Heart Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic heart failure: patients who are diagnosed with chronic heart failure with either preserved or reduced ejection fraction
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study
  Other Names: no intervention

SUMMARY:
The study aims to investigate whether disease progression in patients with chronic heart failure (CHF) can be assessed by new biomarkers, and determine their diagnostic value. The study also intends to describe comparison of echocardiography with cardiopulmonary function test in CHF patients, and relating these cardiac functional parameters to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* with symptoms and signs in NYHA Ⅱ~Ⅳ
* with cardiac structural changes confirmed by echocardiography

Exclusion Criteria:

* with other severe diseases combined and will be alive for less than 12 months
* hard to participate in the investigation or accept the follow-up visits
* pregnant or lactating women
* during the acute phase of ST-elevation acute myocardial infarction, stroke, severe infection and other critical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are diagnosed with chronic heart failure with either preserved or reduced ejection fraction in NYHA Ⅱ~Ⅳ
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-12; Primary Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
main adverse cardiovascular and cerebrovascular events, MACCE | 10 years
  MACCE includes all-cause mortality, cardiovascular mortality, nonfatal myocardial infarction, nonfatal stroke, target lesion revascularization and HF rehospitalization
cardiovascular mortality | 10 years

SECONDARY OUTCOMES:
all-cause mortality | 10 years
new myocardial infarction | 10 years
new stroke | 10 years
heart failure rehospitalization | 10 years
quality of life | 10 years
  described in quality of life scores
worsening of renal function | 10 years
  either an increase of 0.3 mg/dl in serum creatinine or a 20% decrease in eGFR compared with baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided